CLINICAL TRIAL: NCT00468884
Title: Pharmacokinetics and Pharmacodynamic Effects of Oral GLP-1 and PYY3-36: a Proof of Concept Study in Healthy Subjects
Brief Title: Oral Administration of Peptides; Absorption From Gastrointestinal Tract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oral GLP-1 and PYY
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Kinetics of GLP-1 and PYY3-36; increasing oral doses
MeSH Terms: interventions — peptide YY (3-36)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Increasing doses of GLP-1
Drug: PYY3-36

SUMMARY:
Context: Oral formulations of GLP-1 and PYY3-36, two satiety peptides, were studied. An oral delivery system would be preferable in many of the possible therapeutic indications of these peptides.

Objectives: Our objective was to establish the pharmacological profile of increasing oral doses of GLP-1 and PYY3-36 in healthy volunteers. In addition, the pharmacological effects of GLP-1 were investigated.

Setting: Single center escalating dose study with oral applications. Subjects and Methods: In the first part, GLP-1 was given orally to 6 male subjects; the treatment consisted of one of the following oral doses of either GLP-1 (0.5, 1.0, 2.0 and 4.0 mg) or placebo. In the second part, PYY3-36 was given orally to another 6 healthy male subjects; the treatment consisted of one of the following oral doses of either PYY3-36 (0.25, 0.5, 1.0, 2.0 and 4.0 mg) or placebo.

DETAILED DESCRIPTION:
The study was conducted as a phase I, open, placebo-controlled, dose-escalating study. In part I, six treatments, separated by at least 7 days, were performed in 6 male subjects; treatments consisted of one oral dose of GLP-1(7-36 amide) (0.5, 1.0, 2.0, and 4 mg) or placebo; the last treatment was an intravenous infusion of GLP-1 given for 45 min (0.4 pmol/kg per min infused for 45 min). The treatments were identical in design except for the oral dose of GLP-1. In part II, six oral treatments, separated by at least 7 days, were given in an additional 6 male subjects; treatments consisted of one oral dose of PYY3-36 (0.25, 0.5, 1.0, 2.0, and 4 mg) or placebo; an intravenous infusion of PYY3-36 could not be given as no GMP conform PYY3-36 was available for use in humans. Blood was drawn in regular intervals in EDTA tubes containing aprotinin (500 kIU/ml blood) and a DPP-IV inhibitor for hormone determinations: -30, -15, 0, 15, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300 min.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* females

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of GLP-1 and PYY3-36

SECONDARY OUTCOMES:
Effect on ghrelin secretion
Effect on insulin (GLP-1 only)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital, 4031 Basel, Switzerland
Locations (1):
- Clinical Research Centre, University Hospital, Basel, Switzerland

REFERENCES:
- [Background] Degen L, Oesch S, Casanova M, Graf S, Ketterer S, Drewe J, Beglinger C. Effect of peptide YY3-36 on food intake in humans. Gastroenterology. 2005 Nov;129(5):1430-6. doi: 10.1053/j.gastro.2005.09.001. PMID 16285944